CLINICAL TRIAL: NCT03604640
Title: Physical Training and Health Education in the Prevention of Hospital-associated Functional Impairment in Elderly Patients
Brief Title: Physical Training and Health Education in Hospitalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Jose Antonio SERRA-REXACH (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Jose Antonio SERRA-REXACH, Head Of Geriatry Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGECAR PLUS
Record Dates: First submitted 2018-06-28; First posted 2018-07-27 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Functionally-Impaired Elderly
Keywords: Functional impairment; Hospital associated disability
MeSH Terms: interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention)
- Physical and educational program (Experimental)
  Interventions: Other: Physical Training

INTERVENTIONS:
Other: Physical Training — Physical exercise program and health education
  Arms: Physical and educational program

SUMMARY:
The Activity in GEriatric acute CARe (AGECAR) Plus Health Education is a randomized control trial to assess the effectiveness of an intrahospital exercise and health education program during short hospital stays for improving functional capacity of patients aged 75 years or older.

DETAILED DESCRIPTION:
This research aims to investigate the effect of a training program using gait and muscle training and health education, over the functional capacity of elderly hospitalized patients.

The Randomized controlled trial with patients hospitalized in the Acute Care Unit of the Geriatric Department. Participants aged 75 years or older admitted for a short hospital stay will be randomly assigned in a four-week block, to either usual care (control) group or an intervention (training group). Participants allocated in the control group will receive standard hospital care. Participants allocated in the intervention group will perform during hospitalization, training program (30 minutes per session, two sessions per day, lower limb strength training, balance training, walking and inspiratory muscle training) and also health education. Health education consists of several informational activities. Each activity session will teach the patient and caregiver how to perform the exercises to ensure they will continue to be performed at home and before discharge the entire session will be devoted to reviewing the entire program. The type, frequency and progression of the exercises to be carried out will be reviewed; they will be explained how to do them at home and given personalized written instructions with illustrations of the exercises. Also, after one month and two months of discharge, the professional with whom they have completed the training will call them to insist on the completion of the program or to clarify any doubts that may exist.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include people aged 75 years or older recruited from patients admitted into the Geriatrics Department of the Hospital General Universitario Gregorio Marañón (Madrid, Spain).
* Able to ambulate, with or without personal/technical assistance.
* Able to communicate.
* Informed consent: Must be capable and willing to provide consent.

Exclusion Criteria:

* Duration of hospitalization < 72 hours
* Any factor is precluding performance of the physical training program or testing procedures as determined by the attending physician. These factors include, but are not limited to the following:
* Terminal illness.
* Not capable of ambulation.
* Unstable cardiovascular disease or other medical condition.
* Severe dementia.
* Unwillingness to either complete the study requirements or to be randomized into control or intervention group.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 260 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recover basal functional capacity | Three months after discharge
  Changes in the number of Activities of daily living (ADLs) that the patients could perform independently. The six basic ADLs include: bathing, dressing, toileting, transferring, continence, and eating. For each ADL, a score of 0 is assigned for dependence and 1 for independence. A summary scale is constructed by summing the individual ADLs (range of 0-6). Recovery is defined as performance that is at least as good at discharge or 3-months postdischarge as it was at baseline.

SECONDARY OUTCOMES:
Recover basal functional status by Barthel Index of Activities of Daily Living | Three months after discharge
  Change in functional status as measured by other scale of physical function: Barthel Index. This index measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL). Including: feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing. Scoring 0 points would be dependent in all assessed activities of daily living, whereas a score of 100 would reflect independence in these activities. Low scores on individual items highlight areas of need. Recovery is defined as performance that is at least as good at discharge or 3-months postdischarge as it was at baseline.
Ability to walk independently | Three months after discharge
  Changes in functional Ambulation Classification (FAC) scale as one of five functional levels of ambulation (range of 0-4). A score of 0 is assigned if the patient cannot walk, one if the patient requires continuous manual contact to support the body, 2 for light or intermittent manual contact to assist balance, 3 for independent but supervised ambulation, and 4 for independent ambulation on level surfaces or stairs. Recovery is defined as performance that is at least as good at discharge or 3-months postdischarge as it was at baseline.
Physical capacity by the Short Physical Performance Battery (SPPB) | Measurements are taken on the day of admission to the study and the day of discharge from the hospital, an average of 6 days of hospital stay.
  Changes in functional status as measured by the Short Physical Performance Battery (SPPB). SPPB is measured at admission and discharge. Consists of 3 components: standing balance, gait speed, and repeated chair rise. Balance includes standing with feet side-by-side, semi-tandem, and tandem stance. Gait speed scores reflected the time needed to walk 4 m. Repeated chair rise is scored based on time to complete 5 chair rises. Each SPPB component is scored from 0 to 4, and the total sore ranged was 0-12 with higher scores indicating better function. Recovery is defined as performance that is at least as good at discharge as it was at baseline.
Physical capacity by the Alusti test | Measurements are taken on the day of admission to the study and the day of discharge from the hospital, an average of 6 days of hospital stay.
  Changes in functional status as measured by the by the Alusti test. The Alusti test is built in its two versions, complete and abbreviated with below variables: 1) Passive joint mobility 2) Active muscle mobility 3) Transfer from decubitus-supine to seat 4) Sitting trunk 5) Transfer from sitting to standing 6) Standing 7) Walk 8) Operating range 9) Tandem with closed eyes 10) Monopodal support with closed eyes. Each of the variables has a score ranging from 0 to 2, 5, 7, 10 and 25 thresholds. The maximum score that can be obtained in the full Alusti test is 100 points and in the short version of 50: they correspond, respectively, to a situation of excellent/preserved mobility. The minimum score for both versions is 0 points, which would correspond to a total dependency situation. Recovery is defined as performance that is at least as good at discharge as it was at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Serra, PhD, Principal Investigator — HGU Gregorio Marañon
Locations (1):
- Hospital general Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez-Lopez C, Mayordomo-Cava J, Zarralanga-Lasobras T, Romero-Estarlich V, Vidan MT, Ortiz-Alonso J, Valenzuela PL, Rodriguez-Romo G, Lucia A, Serra-Rexach JA. Exercise Intervention and Hospital-Associated Disability: A Nonrandomized Controlled Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2355103. doi: 10.1001/jamanetworkopen.2023.55103. PMID 38329757